CLINICAL TRIAL: NCT02346058
Title: Evaluate the Efficacy and Safety of Esarin Gel in the Treatment of Chronic Venous Insufficiency or Varicose Vein Combine With Superficial Vein Thrombophlebitis in Outpatient
Brief Title: Efficacy and Safety of Esarin Gel in Chronic Venous Insufficiency and Varicose Veins
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ten Sun Pharma Company Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SF13136A
Record Dates: First submitted 2015-01-13; First posted 2015-01-26 (Estimated); Last update posted 2015-01-26 (Estimated); Status verified 2013-06

CONDITIONS: Chronic Venous Insufficiency; Varicose Vein; Superficial Vein Thrombophlebitis
MeSH Terms: conditions — Varicose Veins

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Esarin Gel (Experimental): Dosage form:One tube of Esarin Gel contains 20 gm of compound. Each gm contains:10 mg Heparinoid, 10 mg Escin, 50 mg Diethylamine Salicylate.
  Dosage and frequency: Approx. 3-5 cm Gel was applied topically on skin.twice daily.
  Duration: 28 days.
  Interventions: Drug: Esarin Gel

INTERVENTIONS:
Drug: Esarin Gel

SUMMARY:
Evaluation efficacy and safety of Esarin Gel in subjects with chronic venous insufficiency or varicose veins combine superficial vein thrombophlebitis.

DETAILED DESCRIPTION:
Open-label,non-controlled study design with three visits (pre-treatment/baseline, treatment day 14 and day 28). Administered Esarin Gel twice daily for 28 days in subjects with chronic venous insufficiency rated between CEAP 0 and 3 or varicose veins combine superficial vein thrombophlebitis, in comparison to the pre-treatment.

ELIGIBILITY:
1. Inclusion Criteria:

   * Patients of both sexes, aged above 20 years old.
   * The patient has confirmed his/her willingness to participate in the study, after being informed about all the aspects of the study that might be relevant for his/her decision to participate, and has signed and dated the informed consent form, as approved by the Institutional Review Board/ Ethics Committee (IRB/EC).
   * Presence of chronic venous insufficiency which is rated between functional classes CEAP 0 and 3.(CEAP Classes: C0:no visible or palpable signs of venous disease, C1:telangiectasies or reticular veins. C2 :apparent Varicose veins, C3 :Edema)
   * Diagnosed with superficial vein thrombophlebitis and have skin reaction by redness, swelling, fever and pain symptoms.
2. Exclusion Criteria:

   * Known allergy to the product's ingredients
   * pregnant or breastfeeding
   * patient is joining to any other clinical trail
   * Patient has not sign the informed consent form
   * Deep vein thrombosis
   * Cellulitis
   * Stasis dermatitis
   * The patient is taking non-steroids anti-inflammatory drugs( include oral ,topical creams or patch form)

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2013-10; Primary Completion 2014-06 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Change in subject's leg swelling | 28 days
  Change from pre-treatment (baseline) in the thigh circumference on treatment day 14 and day 28. Using the tape measure to measure the thigh circumference.
Change in subject's leg pain | 28 days
  Change from pre-treatment (baseline) in subject's leg pain on treatment day 14 and day 28. For the assessment of pain, a numerical rating scale (0-10; 0(zero) meaning "no pain" and 10 (ten) "the worst pain") is used.

SECONDARY OUTCOMES:
Safety Assessment through the adverse events reports | 28 days
Improvement of patient's quality of life | 28 days
  Improvement of patient's general activities, mood and sleeping from pre-treatment (baseline) to day 14 and day 28 during Esarin Gel treatment period.

CONTACTS AND LOCATIONS:
Overall Officials: Chung C. Wang, Principal Investigator — Taichung Veterans General Hospital
Locations (1):
- Taichung Veterans General Hospital, Taichung, Taichung, Taiwan